CLINICAL TRIAL: NCT05886270
Title: Implementation of the Child Housing Assessment for a Safe Environment
Acronym: CHASE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Green and Healthy Homes Initiative (Unknown); US Department of Housing and Urban Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MDHHU0059-20; IRB00018899 (Other: JHSPH IRB)
Record Dates: First submitted 2022-08-04; First posted 2023-06-02 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Accident Injury; Home Injury
MeSH Terms: conditions — Accidental Injuries

STUDY DESIGN:
Intervention Model Description: A total of 300 homes in Baltimore City and Baltimore County will be studied, which will be referred from two of GHHI's currently active programs, DSS Foster Care Homes Program (FCHP, n=200 homes) and Amerigroup Maryland Asthma Program (AMAP, n=100 homes), which are Medicaid eligible children referred from Amerigroup-Maryland into GHHI's asthma home-visiting program. The investigators selected families in FCHP and AMAP because they are a representative and generalizable population of low-income children known to have a greater risk of home injuries.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants (Experimental): This arm consists of 300 homes of low-income families with children < 7 years of age who are referred from two of GHHI's currently active programs, DSS Foster Care Homes Program, and Amerigroup Maryland Asthma Program.
  Interventions: Other: Housing Assessment/Safety Modifications

INTERVENTIONS:
Other: Housing Assessment/Safety Modifications — A GHHI Assessor will complete three home visits to assess home injury hazards and provide a scope of work that includes home modifications that directly address each of the identified home injury hazards. The Assessor will also provide do-it-yourself education materials and injury prevention supplies to assist them in completing the modifications.

SUMMARY:
This implementation study uses a multi-method quantitative and qualitative, non-experimental design to estimate the magnitude of home injury risks, identify strategies for addressing those risks and sustaining those interventions, and to calculate the costs of housing-related modifications to prevent childhood home injuries. The study objectives are to: Aim 1. Implement injury prevention measures based on safety hazards identified using the CHASE Tool within 300 low-income households (at or below 80% AMI) in Baltimore City or County; Aim 2. Determine the costs of the injury prevention measures completed by residents and/or professional providers; Aim 3. Conduct a formative evaluation using mixed methods to 3a. determine feasibility of incorporating injury prevention into residential programs from the perspective of installers and residents, including identifying barriers and facilitators, and 3b. understand the consistency of implementing and maintaining the injury prevention measures across referral sources, by residents and staff.

DETAILED DESCRIPTION:
To address the gap between known preventative factors for child home injuries and the uptake of those prevention approaches by high-risk families, the hazards must be systematically and rigorously assessed, and modifications properly implemented and evaluated. Although there are standardized approaches to assess and address particular home health hazards, such as lead paint, asthma, there is no standard tool for injury control. The study team has developed and tested a tool to assess child injury risks in the home (CHASE Tool). The study team has adapted the existing CHASE tool, found in the article by Shields et al 2019, to specify home modifications needed for 15 priority injury hazards that are the focus of this project based on the literature, availability of prevention measures, and the preliminary studies; they include: scalds, falls, fires, crush/cut/pierce injuries, poisonings, and strangulation) however, the time and cost burden to conduct the assessments on a large scale and to implement evidence-based modifications have not been documented, nor is there information available about residents' willingness to accept these modifications. Thus, the investigators propose to combine the child injury prevention expertise of the Johns Hopkins Center for Injury Research and Policy faculty with the home modification and community outreach expertise of Green and Healthy Homes Initiative (GHHI) to demonstrate a new way to improve the safety of children's homes.

The existing CHASE tool, found in the article by Shields et al 2019, has been adapted to specify home modifications needed for 15 priority injury hazards that are the focus of this project based on the literature, availability of prevention measures, and the preliminary studies; they include: scalds, falls, fires, crush/cut/pierce injuries, poisonings, and strangulation.

This project represents the next step in the CHASE project through which the following objectives will be met: Objective 1. Implement injury prevention measures based on safety hazards identified using the CHASE Tool within 300 low-income households (at or below 80% AMI) in Baltimore City or Baltimore County; Objective 2. Determine the costs of the injury prevention measures completed by residents and/or professional providers; Objective 3. Conduct a formative evaluation using mixed methods to 3a. determine feasibility of incorporating injury prevention into residential programs from the perspective of installers and residents, including identifying barriers and facilitators, and 3b. understand the consistency of implementing and maintaining the injury prevention measures across referral sources, by residents and staff.

The Implementation study will be conducted in five phases including the following. Phase 1: Community Engagement. Phase 2: The Enrollment Phase including an initial home visit and assessment for injury risks, CHASE Family Feedback Form creation and education including guidance about needed modifications. Phase 3: Re-Assessment Phase which includes a second home visit to assess change, perform modifications when needed, and survey to understand barriers and facilitators. Phase 4: Follow-Up to measure sustainability of modifications and obtain feedback on the program. Phase 5: Evaluation and Dissemination of results.

The study will enroll a sample of N=300 homes of low-income families with children < 7 years of age who are referred from two of GHHI's currently active programs, Department of Social Services (DSS) Foster Care Homes Program (FCHP, n=200 homes) and Amerigroup Maryland Asthma Program (AMAP, n=100 homes), which are Medicaid eligible children referred from Amerigroup-Maryland into GHHI's asthma home-visiting program.

In addition to completing the three objectives, a user-friendly CHASE Home Safety Modifications Tool Kit and online training module for utilization by other programs working in homes with children will be created and disseminated, thus expanding the potential impact of the present work and HUD's to other housing service providers and beneficiaries nationally.

ELIGIBILITY:
Inclusion Criteria:

* Parent or guardian (or an emancipated minor who meets all other inclusion criteria) whose household is participating in either the GHHI DSS Foster Care Homes Program (FCHP) OR GHHI Amerigroup Maryland Asthma Program (AMAP)
* Households with at least one child under 7 years of age, or foster care families planning to host a child under 7
* The child under 7 years of age lives with the parent or legal guardian most of the time
* Income at or below 80% AMI as defined by US Department of Housing and Urban Development (HUD)
* A home address in Baltimore City or Baltimore County

Exclusion Criteria:

* Parent or guardian whose household is participating is not in either the GHHI DSS Foster Care Homes Program (FCHP) OR GHHI Amerigroup Maryland Asthma Program (AMAP)
* Household does not have at least one child under 7 years of age, or foster care families are not planning to host a child under 7
* The child under 7 years of age does not live with the parent or legal guardian most of the time
* Income is not at or below 80% AMI as defined by HUD
* The home address is not in Baltimore City or Baltimore County

Max Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2022-06-24 (Actual); Primary Completion 2025-12-05 (Actual); Study Completion 2025-12-05 (Actual)

PRIMARY OUTCOMES:
Change in number of Poison Storage hazards | Baseline, 1 month, 3 months
  Poison storage injury hazards will be identified using the CHASE Tool. Fail criteria include: "Your medicine is not locked up" and "Your household products are not locked up."
Change in number of Smoke Alarms hazards | Baseline, 1 month, 3 months
  Smoke alarm injury hazards will be identified using the CHASE Tool. Fail criteria include: "You do not have a smoke alarm on every level of your home."
Change in number of Fire Escape Safety hazards | Baseline, 1 month, 3 months
  Fire escape safety injury hazards will be identified using the CHASE Tool. Fail criteria include: "You do not have at least two exits in all sleeping areas", "Your fire escape exit (door/window) is not working", and "Your fire escape exit(s) are blocked."
Change in number of Sprinkler System hazards | Baseline, 1 month, 3 months
  Sprinkler system injury hazards will be identified using the CHASE Tool. Fail criteria include: "Your sprinkler system is leaking."
Change in number of Carbon Monoxide Alarm hazards | Baseline, 1 month, 3 months
  Carbon monoxide alarm injury hazards will be identified using the CHASE Tool. Fail criteria include: "You do not have at least one carbon monoxide alarm on each level of the home."
Change in number of Electrical Fire and Shock hazards | Baseline, 1 month, 3 months
  Electrical fire and shock injury hazards will be identified using the CHASE Tool. Fail criteria include: "You have a dangerous power strip", "You have a dangerous electrical cord", "You have wires sticking out", "Your electrical receptacle does not have a cover", "Your electrical receptacle is broken", and "Your electrical breaker is broken."
Change in number of Electrical Tripping Risk hazards | Baseline, 1 month, 3 months
  Electrical tripping injury hazards will be identified using the CHASE Tool. Fail criteria include: "You have electrical extension cords that pose a trip and fall hazard."
Change in number of Hot Water Burn hazards | Baseline, 1 month, 3 months
  Hot water burn injury hazards will be identified using the CHASE Tool. Fail criteria include: "You need to retest the hot water temperature to make sure it is a safe temperature", and "You need a new water heater tank installed."
Change in number of Window Fall hazards | Baseline, 1 month, 3 months
  Window fall injury hazards will be identified using the CHASE Tool. Fail criteria include: "Not all of your windows at or above the second level of the home have window stops or guards."
Change in number of Accidental Strangulation hazards | Baseline, 1 month, 3 months
  Accidental strangulation injury hazards will be identified using the CHASE Tool. Fail criteria include: "Your blinds pose a hazard (you do not have cord protectors or cordless blinds/shades)", and "Your blinds/curtains are not cordless, cord protected, or cord unprotected but inaccessible to the child."
Change in number of Stair Fall hazards | Baseline, 1 month, 3 months .
  Stair fall injury hazards will be identified using the CHASE Tool. Fail criteria include: "Your interior stairs are unsafe", "Your carpet is loose", "Your handrails are defective", and "Your railings are defective."
Change in number of Bathroom Fall hazards | Baseline, 1 month, 3 months
  Bathroom fall injury hazards will be identified using the CHASE Tool. Fail criteria include: "Your shower or tub floor surface needs to be deep cleaned before non-slip decals can be applied", "Your shower or tub floor surface needs to be cleaned before non-slip decals can be applied", "You do not have grab bars in your bath tub(s)/shower(s)", and "You do not have a secured, structurally sound shower door."
Change in number of Protruding Nail hazards | Baseline, 1 month, 3 months
  Protruding nails will be identified using the CHASE Tool. Fail criteria include: "You have nails or screws that stick out of the walls and floors that could hurt someone."
Change in number of Falling Furniture hazards | Baseline, 1 month, 3 months
  Falling furniture injury hazards will be identified using the CHASE Tool. Fail criteria include: "You have an entertainment center(s) > 3 ft. above the ground that is not secured to the wall", "You have a book case in the room that is not secured to the wall", "You have a flat screen TV in the room that is not secured to the wall", "You have a traditional TV in the room that is not secured to the wall", and "You have a stove that is not secured to the wall or cabinet/counter."
Change in number of Stair Gate hazards | Baseline, 1 month, 3 months
  Stair gate injury hazards will be identified using the CHASE Tool. Fail criteria include: "You do not have a stair gate installed at the top or bottom of the stairs on the 2nd, and if applicable, 3rd floor", "Not all the stair gates at the top of the stairs are hardware mounted", and "The basement does not have a stair gate at the bottom of the stairs and the top of the stairs, if there is no door at the top of the stairs."

SECONDARY OUTCOMES:
Cost of installing injury prevention measures | 1 month, 3 months
  Determine the costs of the injury prevention measures completed by residents and/or professional providers.
Change in participants' self-reported rates of experienced barriers and facilitators to incorporating injury prevention tools in their home. | Baseline, 1 month, 3 months
  The Health Belief Model Questionnaire will be used to determine the feasibility of incorporating injury prevention into residential programs. Feasibility will be measured by participants' self-reported rates of experienced barriers and facilitators to incorporating injury prevention tools in their home.
Change in qualitative descriptions of participants' confidence to make and maintain injury prevention measures in their home. | 1 month, 3 months
  The Follow-Up Interview will be used to understand the consistency of implementing and maintaining the injury prevention measures across participants. Consistency will be measured by participants' qualitative descriptions of their confidence to make and maintain the changes.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Shields, PhD, Principal Investigator — Johns Hopkins Center for Injury Research and Policy
Locations (1):
- Johns Hopkins Center for Injury Research & Policy, Baltimore, Maryland, United States